CLINICAL TRIAL: NCT03501797
Title: Efficacy of Choir Singing on Verbal, Cognitive, Emotional, and Neural Recovery From Aphasia
Brief Title: Choir Singing in Aphasia Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Hospital District of Helsinki and Uusimaa (Other); Helsinki-Uusimaa Aphasia and Stroke Association (Unknown); Finnish Brain Association (Unknown); Outloud Ltd (Unknown); University of Barcelona (Other); University of Melbourne (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Teppo Sarkamo, Academy of Finland Research Fellow, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 306625
Record Dates: First submitted 2018-02-16; First posted 2018-04-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early singing intervention (AB) (Experimental): Participants receive a 16 weeks of singing-based rehabilitation and standard care (SC) followed by 16 weeks of SC only.
  Interventions: Behavioral: Singing-based rehabilitation; Other: Standard care
- Late singing intervention (BA) (Experimental): Participants receive a 16 weeks of SC only followed by 16 weeks of singing intervention and SC.
  Interventions: Behavioral: Singing-based rehabilitation; Other: Standard care

INTERVENTIONS:
Behavioral: Singing-based rehabilitation — The singing-based rehabilitation is a combination of group-training (16 weeks, 1 x week, 90 min), which utilizes a novel combination of traditional senior choir singing and singing-based speech training protocols, and home training (16 weeks, ≥ 3 x week, ≥ 30 min) in which the choir material is trained with a tablet computer.
Other: Standard care — Standard care comprises all rehabilitation and care services (e.g. speech therapy, physical and occupational therapy, neuropsychological rehabilitation) received by the patients in the Finnish health care system

SUMMARY:
This study evaluates the verbal, cognitive, emotional, and neural efficacy of a choir singing intervention in chronic aphasic patients and their caregivers. Using a cross-over RCT design, half of the participants receive a 4-month singing intervention during the first half of the study and half of the participants during the second half of the study.

DETAILED DESCRIPTION:
BACKGROUND: Singing is a highly stimulating and versatile activity for the brain, combining vocal-motor, auditory, linguistic, cognitive, emotional, and social brain processes, both in the left and right hemisphere. The capacity to sing is often preserved in aphasia after stroke, and singing-based methods, such as Melodic Intonation Therapy (MIT), can be effective in rehabilitating speech production in aphasics. Also emotionally and socially, singing could provide a powerful alternative channel for aphasic patients to express their emotions and interact with others, but the communal or group-level use of singing in aphasia rehabilitation has not been systematically studied.

AIMS: The purpose of the study is to determine the clinical and neural efficacy of a novel choir singing intervention in subacute/chronic aphasia. Specifically, the targeted outcomes are (i) verbal and vocal-motor skills, (ii) cognitive skills, (iii) emotional functioning and quality of life, (iv) caregiver psychological well-being, and (v) structural and functional neuroplasticity. In addition, the capacity of singing and music learning in aphasia is explored.

METHODS: Subjects are 60 stroke patients with at least minor aphasia (≥ 6 months post-stroke) and their family members (FMs, N = 60) from Helsinki area recruited to a cross-over RCT study. Participants are randomized to two groups [N = 60 in both (30 patients, 30 FMs)], which receive a 16-week choir intervention either during the first (AB group) or second (BA group) half of the follow-up. The intervention is a combination of group training, which utilizes a novel combination of traditional senior choir singing and MIT-like speech training protocols, and home training in which the choir material is trained with a tablet computer. All patients are evaluated at baseline, 5-month, and 9-month stages with language, cognitive, and auditory-music tests and questionnaires. Half of the patients (N = 30) also undergo electroencephalography (EEG) and structural and functional magnetic resonance imaging (s/fMRI). FMs are evaluated with questionnaires.

ELIGIBILITY:
The following inclusion criteria are used in patient recruiment:

1. age over 18
2. Finnish-speaking
3. time since stroke > 6 months
4. at least minor non-fluent aphasia due to stroke (BDAE Aphasia Severity Rating scale score ≤ 4)
5. no hearing deficit
6. no severe cognitive impairment affecting comprehension (the patient is able to understand the purpose of the study and give an informed consent)
7. no neurological / psychiatric co-morbidity or substance abuse
8. ability to produce vocal sound (through singing or humming).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Communication ability | Change from baseline at 5 months and 9 months
  Total score of the Communication Action Log (CAL) questionnaire (range 0-180, higher score indicates better outcome)
Spontaneous speech production | Change from baseline at 5 months and 9 months
  Spontaneous Speech subscale score of the Western Aphasia Battery (WAB) (range 0-20, higher score indicates better outcome)
Connected speech informativeness | Change from baseline at 5 months and 9 months
  Percentage of correct information units (CIUs) produced in a picture description task
Repetition of words and sentences | Change from baseline at 5 months and 9 months
  Repetition subscale score of the Western Aphasia Battery (WAB) (range 0-100, higher score indicates better outcome)
Verbal agility | Change from baseline at 5 months and 9 months
  Verbal Agility subtest score of the Boston Diagnostic Aphasia Examinaton (BDAE) (range 0-14, higher score indicates better outcome)
Naming and word finding | Change from baseline at 5 months and 9 months
  Naming and Word Finding subscale score of the Western Aphasia Battery (WAB) (range 0-100, higher score indicates better outcome)
Verbal comprehension | Change from baseline at 5 months and 9 months
  Sequential Commands subtest score of the Western Aphasia Battery (WAB) (range 0-80, higher score indicates better outcome)

SECONDARY OUTCOMES:
Executive function (correct responses) | Change from baseline at 5 months and 9 months
  Simon Task: score (range 0-100, higher score indicates better outcome)
Executive function (reaction times) | Change from baseline at 5 months and 9 months
  Simon Task: reaction time mean (ms)
Attention (correct responses) | Change from baseline at 5 months and 9 months
  Flexible Attention Test (FAT): score (range 0-48, higher score indicates better outcome)
Attention (reaction times) | Change from baseline at 5 months and 9 months
  Flexible Attention Test (FAT): reaction time mean (ms)
Working memory | Change from baseline at 5 months and 9 months
  Word Span subtest score of the Kielelliset Arviointitehtävät (KAT) (range 0-30, higher score indicates better outcome)
Verbal memory | Change from baseline at 5 months and 9 months
  Logical Memory subtest score of the Wechsler Memory Scale III (WMS-III) (range 0-80, higher score indicates better outcome)
Verbal learning | Change from baseline at 5 months and 9 months
  Word Lists subtest score of the Wechsler Memory Scale III (WMS-III) (range 0-84, higher score indicates better outcome)
Singing ability | Change from baseline at 5 months and 9 months
  Acoustic features (e.g., pitch, rhythm, intensity) analyzed from recorded production of familiar and novel songs using acoustic analysis software
Music perception | Change from baseline at 5 months and 9 months
  Montreal Battery of Evaluation of Amusia (MBEA) score (range 0-30, higher score indicates better outcome)
Functional stroke recovery | Change from baseline at 5 months and 9 months
  Total score of the Stroke Impact Scale (SIS) questionnaire (range 0-900, higher score indicates better outcome)
Depression | Change from baseline at 5 months and 9 months
  Total score of the Center for Epidemiological Studies Depression Scale (CES-D) questionnaire (range 0-60, lower score indicates better outcome)
Mood | Change from baseline at 5 months and 9 months
  Total score of the Visual Analog Mood Scales (VAMS) questionnaire (range 0-800, higher score indicates better outcome)
Social interaction | Change from baseline at 5 months and 9 months
  Total score of the Social Provision Scale (SPS) questionnaire (range 24-96, higher score indicates better outcome)
Caregiver burden | Change from baseline at 5 months and 9 months
  Total score of the Zarit Burden Interview (ZBI-22) questionnaire (range 0-88, lower score indicates better outcome)
Psychological stress of the caregiver | Change from baseline at 5 months and 9 months
  Total score of the General Health Questionnaire (GHQ-12) (range 0-36, lower score indicates better outcome)
Electroencephalography (EEG) | Change from baseline at 5 months and 9 months
  Amplitude and latency of event-related potentials (ERPs) associated with learning and memory in two auditory tasks
Structural magnetic resonance imaging (sMRI): MPRAGE sequence | Change from baseline at 5 months and 9 months
  Grey matter volume in frontotemporal, frontoparietal, and limbic brain regions
Structural magnetic resonance imaging (sMRI): DTI sequence | Change from baseline at 5 months and 9 months
  Structural connectivity of intra- and interhemispheric white matter tracts
Functional magnetic resonance imaging (fMRI): resting-state | Change from baseline at 5 months and 9 months
  resting-state fMRI sequence: functional connectivity of frontotemporal, frontoparietal, and limbic brain networks
Functional magnetic resonance imaging (fMRI): singing-related activity | Change from baseline at 5 months and 9 months
  task-based fMRI sequence: frontotemporal, frontoparietal, and limbic activation patterns associated with the perception, vocal repetition, and recall of novel songs

CONTACTS AND LOCATIONS:
Overall Officials: Teppo Särkämö, PhD, Principal Investigator — University of Helsinki
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Department of Neurology, Rehabilitation Unit, Helsinki
  - Helsinki-Uusimaa Aphasia and Stroke Association, Helsinki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Molina N, Pitkaniemi A, Siponkoski ST, Moisseinen N, Kuusela L, Laitinen S, Sarkamo ER, Pekkola J, Melkas S, Schlaug G, Kleber B, Sihvonen AJ, Sarkamo T. Functional neuroplasticity in chronic post-stroke aphasia following a singing intervention in a cross-over randomised trial. Sci Rep. 2025 Jul 29;15(1):27639. doi: 10.1038/s41598-025-11288-0. PMID 40738917
- [Derived] Siponkoski ST, Pitkaniemi A, Laitinen S, Sarkamo ER, Pentikainen E, Eloranta H, Tuomiranta L, Melkas S, Schlaug G, Sihvonen AJ, Sarkamo T. Efficacy of a multicomponent singing intervention on communication and psychosocial functioning in chronic aphasia: a randomized controlled crossover trial. Brain Commun. 2022 Dec 27;5(1):fcac337. doi: 10.1093/braincomms/fcac337. eCollection 2023. PMID 36687394